CLINICAL TRIAL: NCT01670331
Title: Psychological Preparation Prior to Bariatric Surgery: A Feasibility Study
Brief Title: Psychological Preparation Prior to Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STH16575
Record Dates: First submitted 2012-07-10; First posted 2012-08-22 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Obesity; Psychological Disorders
MeSH Terms: conditions — Obesity; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychological preparation (Active Comparator): Patients undergo 3 seminar sessions with the bariatric psychologist prior to their surgery. These will aim to prepare them for the lifestyle changes that will occur / they will have to make after surgery
  Interventions: Behavioral: Psychological preparation
- Surgery as usual (No Intervention): Patients will proceed to surgery as usual. They will complete psychological assessment forms at their follow up clinic sessions.

INTERVENTIONS:
Behavioral: Psychological preparation — Session 1: Help patients understand their relationship to food. Patients complete a 'food diary' as 'homework'. Give information about lifestyle changes after surgery. Presents the model of 'stress' and how it influences 'overeating', to develop a more balanced lifestyle and better QoL.
  Session 2: 'Intervention' using Compassion Focussed Therapy model to understand relationship to food from their diary. Help develop a 'minimising overeating plan' (a 'relapse prevention' plan). Help learn to meet needs in other ways than food.
  Session 3: Focus on physical body. Current body image, explore hopes and expectations for after surgery. Consider how to manage changes to social reactions and sexual relationships that may occur.
  Other Names: Pre-bariatric surgery psychological programme
  Arms: Psychological preparation

SUMMARY:
Is it feasible to perform a randomized controlled trial to assess whether or not psychological preparation seminars prior to bariatric (weight loss) surgery are beneficial to the investigators patients?

DETAILED DESCRIPTION:
This is a feasibility study, assessing how possible it would be to perform a randomized controlled trial to see if preoperative psychological or mental health problems impacts on length of stay, short and long term health outcomes, weight loss, and if preoperative counseling has any effect.

ELIGIBILITY:
Inclusion Criteria:

* New referrals to the Sheffield Teaching Hospital Bariatric service

Exclusion Criteria:

* Non-English speakers
* Patients that are not fit for bariatric surgery
* Patients that have already seen the bariatric psychologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-03; Primary Completion 2016-06 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Are there increased scores in the BAROS psychometric tests in patients that undergo psychological preparation prior to bariatric surgery, than in those that do not at 12 months? | 12 months
  At 12 months, patients will attend clinic and complete a battery of psychological assessment questionnaires and the results compared to see if there is a quantifiable difference in the quality of life and mental health outcomes of patients that undergo preparation seminars and those that do not.

SECONDARY OUTCOMES:
Are there increased scores in the PHQ-9 psychometric tests in patients that undergo psychological preparation prior to bariatric surgery, than in those that do not at 12 months? | 12 months
  At 12 months, patients will attend clinic and complete a battery of psychological assessment questionnaires and the results compared to see if there is a quantifiable difference in the quality of life and mental health outcomes of patients that undergo preparation seminars and those that do not.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne E Owers, MB/ChB, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust; Adam Saradjian, DClinPsy, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom